CLINICAL TRIAL: NCT05483673
Title: A Comprehensive Study for Analyzing Orthopedic Patient Experience Patterns in Medical Trials
Brief Title: Analyzing Orthopedic Patient Experience Patterns in Medical Trials
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 86809840
Record Dates: First submitted 2022-07-29; First posted 2022-08-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Orthopedic Disorder
Keywords: orthopedic
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical study enrollment has historically been heavily biased toward specific demographics.

Several people will be invited to participate in this study so that it may collect a variety of data about orthopedic clinical trial experiences and identify barriers to participation as well as the causes of participants' failure or withdrawal.

People with orthopedic disorders who are invited to take part in medical research will benefit from the analysis of the data.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been diagnosed with orthopedic disorder
* Patient has self-identified as planning to enroll in an interventional clinical trial
* Patient is 18 years old

Exclusion Criteria:

* ECOG score of 4
* Patient is pregnant
* Inability to perform regular electronic reporting
* Patient does not understand, sign, and return consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Orthopedic disorder patients who are actively considering enrolling in an interventional clinical trial, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of patients who decide to enroll in an orthopedic clinical trial | 3 months
Rate of patients who remain in orthopedic clinical trial to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hollis AC, Davis ET. Understanding the factors that influence patient participation in Orthopaedic Clinical Trials. Int Orthop. 2018 Aug;42(8):1769-1774. doi: 10.1007/s00264-018-3890-2. Epub 2018 Mar 20. PMID 29560527
- [Background] Trippel SB, Bosse MJ, Heck DA, Wright JG. Symposium. How to participate in orthopaedic randomized clinical trials. J Bone Joint Surg Am. 2007 Aug;89(8):1856-64. doi: 10.2106/JBJS.F.01596. No abstract available. PMID 17671026
- [Background] Somerson JS, Bartush KC, Shroff JB, Bhandari M, Zelle BA. Loss to follow-up in orthopaedic clinical trials: a systematic review. Int Orthop. 2016 Nov;40(11):2213-2219. doi: 10.1007/s00264-016-3212-5. Epub 2016 May 3. PMID 27142421

DOCUMENTS (1):
  • Informed Consent Form (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/73/NCT05483673/ICF_000.pdf